CLINICAL TRIAL: NCT02010619
Title: Internet Delivered Cognitive Behavior Therapy for Body Dysmorphic Disorder - a Randomized Controlled Trial
Brief Title: Internet Delivered CBT for Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Associate professor, M.D., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BDD RCT
Record Dates: First submitted 2013-11-18; First posted 2013-12-13 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Body Dysmorphic Disorder; BDD
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cognitive behavior therapy (Experimental)
  Interventions: Behavioral: Cognitive behavior therapy
- Supportive therapy (Active Comparator)
  Interventions: Behavioral: Supportive therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy
  Arms: Cognitive behavior therapy
Behavioral: Supportive therapy
  Arms: Supportive therapy

SUMMARY:
To evaluate if Internet delivered cognitive behavior therapy is an efficacious treatment when compared to a control group consisting of supportive therapy.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* ≥ 18 years
* primary diagnosis of BDD according to the DSM-5
* BDD-YBOCS ≥20
* regular access to a computer with Internet access and skills to use the web.

Exclusion Criteria:

* psychotropic medication changes within two months prior to the treatment,
* completed CBT for BDD within the last 12 months,
* other primary axis I diagnosis
* current substance dependence
* lifetime bipolar disorder or psychosis
* suicidal ideation
* Axis II diagnosis that could jeopardize treatment participation,
* other current psychological treatment that could affect BDD symptoms
* A serious medical illness that precludes participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Body Dysmorphic Disorder Modification of the Y-BOCS (BDD-YBOCS) | Change in BDD-YBOCS from baseline (week 0) to post-treatment (week 12)

SECONDARY OUTCOMES:
The Montgomery Åsberg Depression Rating Scale - self report (MADRS-S) | Change in MADRS-S from baseline (week 0) to post-treatment (week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst, Stockholm, Huddinge, Sweden

REFERENCES:
- [Result] Enander J, Andersson E, Mataix-Cols D, Lichtenstein L, Alstrom K, Andersson G, Ljotsson B, Ruck C. Therapist guided internet based cognitive behavioural therapy for body dysmorphic disorder: single blind randomised controlled trial. BMJ. 2016 Feb 2;352:i241. doi: 10.1136/bmj.i241. PMID 26837684
- [Derived] Flygare O, Andersson E, Glimsdal G, Mataix-Cols D, Pascal D, Ruck C, Enander J. Cost-effectiveness of internet-delivered cognitive behaviour therapy for body dysmorphic disorder: Results from a randomised controlled trial. Internet Interv. 2023 Jan 24;31:100604. doi: 10.1016/j.invent.2023.100604. eCollection 2023 Mar. PMID 36756354
- [Derived] Flygare O, Enander J, Andersson E, Ljotsson B, Ivanov VZ, Mataix-Cols D, Ruck C. Predictors of remission from body dysmorphic disorder after internet-delivered cognitive behavior therapy: a machine learning approach. BMC Psychiatry. 2020 May 19;20(1):247. doi: 10.1186/s12888-020-02655-4. PMID 32429939
- [Derived] Enander J, Ljotsson B, Anderhell L, Runeborg M, Flygare O, Cottman O, Andersson E, Dahlen S, Lichtenstein L, Ivanov VZ, Mataix-Cols D, Ruck C. Long-term outcome of therapist-guided internet-based cognitive behavioural therapy for body dysmorphic disorder (BDD-NET): a naturalistic 2-year follow-up after a randomised controlled trial. BMJ Open. 2019 Jan 15;9(1):e024307. doi: 10.1136/bmjopen-2018-024307. PMID 30647044